CLINICAL TRIAL: NCT01273376
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group, Phase 2 Study of RX-10100 in Subjects With Major Depressive Disorder.
Brief Title: Safety and Efficacy of RX-10100 to Treat Major Depressive Disorder
Acronym: MDD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rexahn Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010MDD01
Record Dates: First submitted 2011-01-06; First posted 2011-01-10 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Major Depressive Disorder
Keywords: MDD; Depression; Major Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — RX-10100

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- RX-10100 high dose (Experimental): RX-10100
  Study drug is to be given orally, in tablet form, twice daily, for 8 weeks
  Interventions: Drug: RX-10100
- RX-10100 low dose (Experimental): RX-10100
  Study drug is to be given orally, in tablet form, twice daily, for 8 weeks
  Interventions: Drug: RX-10100
- Placebo (Placebo Comparator): Matching placebo is to be given orally, in tablet form, twice daily, for 8 weeks
  Interventions: Drug: RX-10100

INTERVENTIONS:
Drug: RX-10100 — Extended-release tablet, taken twice daily for 8 weeks
  Other Names: Serdaxin®

SUMMARY:
The purpose of this study is to determine whether RX-10100 are effective in the treatment of Major Depressive Disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

• Moderate to severe MDD as determined by the DSM-IV-TR Axis 1 Disorders and by the Montgomery Asberg Depression Rating Scale (MADRS).

Exclusion Criteria:

* Women who are pregnant, women who will be breastfeeding during the study, and women with childbearing potential who are not willing to practice a reliable method of birth control
* Depressive episode duration of less than 1 month
* Lifetime history of any psychotic disorders
* Anxiety disorders
* Significant suicidality
* Clinically significant medical conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2010-12; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Montgomery-Asberg Depression Rating Scale (MADRS)at week 9 | 8 weeks

SECONDARY OUTCOMES:
Change from baseline in Montgomery-Asberg Depression Rating Scale (MADRS) at weeks 3, 5, and 7 | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christine Peterson, Ph.D, Study Director — Rexahn Pharmaceuticals, Inc.
Locations (44):
- United States (44):
  - Rexahn Investigative Site, Cerritos, California
  - Rexahn Investigative Site, Escondido, California
  - Rexahn Investigative Site, Los Angeles, California
  - Rexahn Investigative Site, National City, California
  - Rexahn Investigative Site, Oceanside, California
  - Rexahn Investigative Site, Orange, California
  - Rexahn Investigative Site, San Diego, California
  - Rexahn Investigative Site, Denver, Colorado
  - Rexahn Investigative Site, Brooksville, Florida
  - Rexahn Investigative Site, Gainesville, Florida
  - Rexahn Investigative Site, Jacksonville, Florida
  - Rexahn Investigative Site, Miami Beach, Florida
  - Rexahn Investigative Site, Orlando, Florida
  - Rexahn Investigative Site, St. Petersburg, Florida
  - Rexahn Investigative Site, Tampa, Florida
  - Rexahn Investigative Site -2, Atlanta, Georgia
  - Rexahn Investigative Site, Atlanta, Georgia
  - Rexahn Investigative Site, Oak Brook, Illinois
  - Rexahn Investigative Site, Vernon Hills, Illinois
  - Rexahn Investigative Site, Owensboro, Kentucky
  - Rexahn Investigative Site, Novi, Michigan
  - Rexahn Investigative Site, Las Vegas, Nevada
  - Rexahn Investigative site, Cherry Hill, New Jersey
  - Rexahn Investigative Site, Albuquerque, New Mexico
  - Rexahn Investigative Site, Fresh Meadows, New York
  - Rexahn Investigative Site, New York, New York
  - Rexahn Investigative Site, Cincinnati, Ohio
  - Rexahn Investigative site, Garfield Heights, Ohio
  - Rexahn Investigative Site, Oklahoma City, Oklahoma
  - Rexahn Investigative site, Allentown, Pennsylvania
  - Rexahn Investigative Site, Media, Pennsylvania
  - Rexahn Investigative Site, Scranton, Pennsylvania
  - Rexahn Investigative Site, Anderson, South Carolina
  - Rexahn Investigative Site, Memphis, Tennessee
  - Rexahn Investigative Site, Austin, Texas
  - Rexahn Investigative site, Dallas, Texas
  - Rexahn Investigative Site, Dallas, Texas
  - Rexahn Investigative Sites, Lake Jackson, Texas
  - Rexahn Investigative Site, San Antonio, Texas
  - Rexahn Investigative Site, The Woodlands, Texas
  - Rexahn Investigative Site, Orem, Utah
  - Rexahn Investigative Site, Richmond, Virginia
  - Rexahn Investigative Site (2), Bellevue, Washington
  - Rexahn Investigative Site, Bellevue, Washington